CLINICAL TRIAL: NCT04135859
Title: Physical Activity Lifestyle Intervention for Young Adults With Congenital Heart Disease
Brief Title: Young Adult Congenital Heart Disease Physical Activity Lifestyle Study (YACHD-PALS)
Acronym: YACHD-PALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jamie Jackson (Other)
Responsible Party: Sponsor-Investigator, Jamie Jackson, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB1600717
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiovascular Disease Other; Physical Activity
Keywords: congenital heart disease; physical activity
MeSH Terms: conditions — Motor Activity; Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: Study includes 2 possible conditions to which participants are randomized: (1) Fitbit only and (2) Fitbit + coaching sessions.
Masking Description: Investigator, research assistants, coaches (interventionists), and participants do not know which condition a participant is in until the condition is revealed (opening an envelope with the condition listed) after the participant consents to Phase 2. Envelopes with the conditions were prepared by the study statistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fitbit Only (Active Comparator): In the Fitbit Only arm, participants will receive their exercise prescription, as devised from their baseline exercise stress test results, and a Fitbit. They will undergo a 9 week (interim) and a 22 week assessment (follow-up).
  Interventions: Behavioral: Physical Activity Monitoring
- Fitbit + Coaching Sessions (Experimental): In the Fitbit + Coaching Sessions arm, participants will receive their exercise prescription, as devised from their baseline exercise stress test results, a Fitbit, and will have 8 sessions with a coach (interventionist) over the course of 20 weeks. They will undergo a 9 week (interim) and a 22 week assessment (follow-up).
  Interventions: Behavioral: Physical Activity Lifestyle Intervention; Behavioral: Physical Activity Monitoring

INTERVENTIONS:
Behavioral: Physical Activity Lifestyle Intervention — Coaches work with participants on three elements of behaviors change: (1) changing attitudes towards physical activity; (2) increase perceptions of other people's approval of physical activity for the participants; (3) increase perceptions of control over being physically active. These elements will be delivered using a non-judgmental stance accompanied by promoting appropriate goal-setting.
  Arms: Fitbit + Coaching Sessions
Behavioral: Physical Activity Monitoring — A physical activity monitor (Fitbit) will be provided to both groups.
  Other Names: Fitbit

SUMMARY:
This study will adapt a physical activity lifestyle intervention to emerging adult congenital heart disease (CHD) survivors with the primary goal of increasing physical activity levels.

The study will be split into 2 phases. In Phase 1, participants will be asked to complete questionnaires, wear an accelerometer around the waist for 7 days, and undergo an exercise stress test. The accelerometer and exercise stress test will be used to determine whether participants are eligible to be randomized for the intervention study. In Phase 2, participants will be randomized to one of two conditions: 1) receiving a physical activity tracker (a Fitbit) or 2) receiving a Fitbit AND engaging in videoconferencing sessions with a physical activity coach. During Phase 2, participants will also be asked to complete 3 assessments (weeks 9 and 22, and a 6-month follow-up). The week 9 assessment will consist of completing questionnaires and wearing an accelerometer for 7 days. Week 22 will be similar to week 9 with the addition of a final exercise stress test. The 6-month follow-up will mirror the week 9 assessment.

Participants who are randomized to the videoconferencing condition will be asked to meet with a physical activity coach 8 times over the course of 20 weeks. Coaches will help participants to (1) change attitudes toward physical activity, (2) increase perception of others' approval of physical activity (e.g., family members, peers), and (3) increase participants' perceived control by troubleshooting barriers and increasing efficacy for physical activity. Coaches will use the Fitbit to facilitate self-monitoring and goal setting. Participants in the intervention arm will be asked to participate in a focus group at the conclusion of the study to share their experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18-25 (if 18, must no longer be in high school and no longer living at home)
2. Are diagnosed with moderate or complex structural congenital heart disease
3. Live within 120 miles of Nationwide Children's Hospital

Exclusion Criteria:

1. Do no speak or write proficiently in English
2. Have cognitive impairments that would interfere with the completion of study procedures
3. Are diagnosed with a genetic syndrome (e.g., Downs, Marfans)
4. Have been engaged in a formal exercise program within the past 6 months
5. Underwent open-heart surgery or have had a transcatheter valve replacement in the last 3 months
6. Are otherwise prohibited by their cardiologist to engage in at least moderate levels of physical activity
7. Are unable to complete a treadmill-based exercise stress test
8. Are currently pregnant
9. Have contraindications for exercise based on an exercise stress test (e.g., exercise-induced arrhythmias or evidence of cardiac ischemia)
10. >150 min/weekday of moderate-to-vigorous physical activity per the accelerometer
11. Do not have access or a device for videoconferencing with the coach

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams CA, Wadey C, Pieles G, Stuart G, Taylor RS, Long L. Physical activity interventions for people with congenital heart disease. Cochrane Database Syst Rev. 2020 Oct 28;10(10):CD013400. doi: 10.1002/14651858.CD013400.pub2. PMID 33112424

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fitbit Only | Fitbit + Coaching Sessions
Started | 19 | 17
Completed | 14 | 10
Not Completed | 5 | 7
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal due to screening failure | 1 | 2
Not completed — Did not complete stress test | 3 | 3
Not completed — Did not wear accelerometer and did not complete stress test | 0 | 2

BASELINE CHARACTERISTICS:
Population: Three withdrawn participants (2 from Fitbit + Coaching Sessions arm and 1 from Fitbit Only arm) are excluded from the baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Fitbit Only | Fitbit + Coaching Sessions | Total
Number analyzed (Participants) | 18 | 15 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.2 (1.9) | 22.3 (2.3) | 22.2 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 18 | 14 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 15 | 33
MVPA [Mean (Standard Deviation); unit: Average min/day] | 7.5 (4.8) | 9.4 (5.0) | 8.4 (4.9)
Sedentary Behavior [Mean (Standard Deviation); unit: Average min/day] | 561.2 (100.0) | 580.3 (118.7) | 570.2 (107.8)
VO2Peak [Mean (Standard Deviation); unit: mL/kg/min] | 30.3 (7.1) | 31.4 (8.6) | 30.9 (7.7)

OUTCOME MEASURES:

1. Primary Outcome: Moderate to Vigorous Physical Activity (MVPA)
Description: Baseline to follow-up change in number of minutes spent in moderate to vigorous physical activity as measured by an accelerometer
Time Frame: From baseline to follow-up (approximately 22 weeks).
Population: Two participants in the Fitbit + Coaching group had missing MVPA data
Measure: Mean (Standard Deviation); unit: Average change in minutes per day
Arm/Group | Fitbit Only | Fitbit + Coaching Sessions
Number analyzed (Participants) | 17 | 13
Average change in minutes per day | -0.7 (6.6) | 8.8 (15.7)
Statistical Analysis 1: Comparison: Fitbit Only vs Fitbit + Coaching Sessions; Test type: Superiority; p = .023, Mixed Models Analysis; Mean Difference (Final Values) = 10.3

2. Secondary Outcome: Sedentary Behavior
Description: Baseline to follow-up change in number of minutes spent being sedentary as measured by an accelerometer.
Time Frame: From baseline to follow-up (approximately 22 weeks).
Population: Three participants in the Fitbit + Coaching group had missing data for sedentary behavior
Measure: Mean (Standard Deviation); unit: Average change in minutes per day
Arm/Group | Fitbit Only | Fitbit + Coaching Sessions
Number analyzed (Participants) | 17 | 12
Average change in minutes per day | 13.6 (88.7) | -49.8 (92.3)
Statistical Analysis 1: Comparison: Fitbit Only vs Fitbit + Coaching Sessions; Test type: Superiority; p = .06, Mixed Models Analysis; Mean Difference (Final Values) = -59.0

3. Secondary Outcome: Exercise Tolerance
Description: Baseline to follow-up change in maximal oxygen utilization during physical activity as measured by VO2peak during an exercise stress test.
Time Frame: From baseline to follow-up (approximately 22 weeks).
Population: Three participants from the Fitbit Only group and four participants from the Fitbit + Coaching Sessions group had missing data for VO2peak.
Measure: Mean (Standard Deviation); unit: Average change in mL/kg/min
Arm/Group | Fitbit Only | Fitbit + Coaching Sessions
Number analyzed (Participants) | 14 | 9
Average change in mL/kg/min | 0.41 (2.33) | -0.32 (1.68)
Statistical Analysis 1: Comparison: Fitbit Only vs Fitbit + Coaching Sessions; Test type: Superiority; p = .43, Mixed Models Analysis; Mean Difference (Final Values) = -0.76

ADVERSE EVENTS:
Time Frame: Randomization to follow-up (approximately 22 weeks)
Description: An adverse event is an unanticipated change in cardiovascular, musculoskeletal, or emotional symptoms that are (1) concerning to the participant and (2) results in seeking medical attention, if cardiovascular or musculoskeletal in nature. Any condition that is present at the time that the participant is screened will be considered as baseline and not reported as an adverse event.
Arm/Group | Fitbit Only | Fitbit + Coaching Sessions
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 1/19 | 0/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fitbit Only (N=19) | Fitbit + Coaching Sessions (N=17)
Ankle sprain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Severity: Moderate Relatedness: Unrelated Expectedness: Unexpected

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04135859/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT04135859/ICF_000.pdf